CLINICAL TRIAL: NCT05314959
Title: Physician Awareness of Patients' Preferred Level of Involvement in Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Thythy Pham, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 215830
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Preferred Level of Involvement in Decision Making

STUDY DESIGN:
Intervention Model Description: Women will be randomly assigned to physician awareness or treatment as usual (control) using a 1:1 allocation
Who Masked: Participant
Masking Description: The control group will have usual care, meaning that the physician will NOT see the patient's survey results. The patient is blinded to randomization and will not know whether or not the physician is aware of their preferred level of shared decision making.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician Awareness (Experimental): The physician will have access to the pre-visit Control Preference Scale survey results for women assigned to this group
  Interventions: Other: Physician Awareness
- Usual Care (Active Comparator): The physician will not have access to the pre-visit Control Preference Scale survey results for women assigned to this group
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Physician Awareness — The patients' pre-visit Control Preference Scale responses are shared with their physician.
  Arms: Physician Awareness
Other: Usual Care — The patients' pre-visit Control Preference Scale responses are not shared with their physician.
  Arms: Usual Care

SUMMARY:
Understanding a patient's decision-making preferences can help physicians meet their expectations and may increase patient satisfaction with the decision-making process.

DETAILED DESCRIPTION:
Many health systems are shifting policies to promote greater patient involvement in healthcare delivery. Studies have shown that general medical patients who are more active in their care are more satisfied, more committed, have a better understanding of treatment plans, and experience greater improvements in health and patient-centered outcomes when compared to more passive patients. That being said, studies have found that patients have varying preferences when it comes to decision making. Understanding a patient's decision-making preferences can help physicians meet their expectations and may increase patient satisfaction with the decision-making process.

This awareness of decision-making preferences could be beneficial in treating quality of life conditions. Patients seeking care for pelvic floor disorders make medical decisions aimed toward improving symptoms, function, and quality of life. In a recent study, researchers found that 50% of women preferred active involvement, 45% collaborative and 5% passive. However, patients were 1.56 (95% CI:1.06-2.29) times more likely to report collaborative or passive involvement after their visit (p=0.02) with 40% of patients rating their actual role as active, 48% as collaborative, and 11% as passive. In this study, 37% of women did not experience their preferred level of decision-making. Other studies have similar findings with reported 20-40% discordance between patients' preferred involvement and what was achieved.

Discordance can negatively impact patients' outcomes and experiences of care. Interventions to minimize discordance between patients' preferred and perceived involvement in decision-making may significantly improve their overall experience and satisfaction. One possible intervention is eliciting women's preferred level of involvement in decision making prior to the visit and making this information available to the physician. The current study aims to determine whether physicians' awareness of patients' preferred involvement in decision making prior to their initial urogynecologist visit affects patients' perceived involvement in decision making after their visit.

ELIGIBILITY:
Inclusion Criteria:

* Present to Loyola's Urogynecology clinic for their initial evaluation
* Agree to complete the study questionnaires
* Must be at least 18 years of age
* Must be able to read, speak and write in English

Exclusion Criteria:

* Established patients at Loyola's Urogynecology clinic
* Unable to complete the study questionnaires
* Less than 18 years of age
* Unable to read, speak and write in English

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Discordance rate for the Control Preference Scale | 1 day visit
  The Control Preference Scale assesses patients' preferences for involvement in decision-making. The scale ranks patients' preferences for involvement in their healthcare as either active, collaborative, or passive. Patients' CPS responses will be compared between the intervention and usual care cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Thythy Pham, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crawford MJ, Rutter D, Manley C, Weaver T, Bhui K, Fulop N, Tyrer P. Systematic review of involving patients in the planning and development of health care. BMJ. 2002 Nov 30;325(7375):1263. doi: 10.1136/bmj.325.7375.1263. PMID 12458240
- [Background] Hubbard G, Kidd L, Donaghy E. Preferences for involvement in treatment decision making of patients with cancer: a review of the literature. Eur J Oncol Nurs. 2008 Sep;12(4):299-318. doi: 10.1016/j.ejon.2008.03.004. Epub 2008 May 16. PMID 18486552
- [Background] Sung VW, Raker CA, Myers DL, Clark MA. Treatment decision-making and information-seeking preferences in women with pelvic floor disorders. Int Urogynecol J. 2010 Sep;21(9):1071-8. doi: 10.1007/s00192-010-1155-8. Epub 2010 Apr 28. PMID 20424822
- [Background] Beaver K, Bogg J, Luker KA. Decision-making role preferences and information needs: a comparison of colorectal and breast cancer. Health Expect. 1999 Dec;2(4):266-276. doi: 10.1046/j.1369-6513.1999.00066.x. PMID 11281903
- [Background] Degner LF, Sloan JA. Decision making during serious illness: what role do patients really want to play? J Clin Epidemiol. 1992 Sep;45(9):941-50. doi: 10.1016/0895-4356(92)90110-9. PMID 1432023
- [Background] Tariman JD, Berry DL, Cochrane B, Doorenbos A, Schepp K. Preferred and actual participation roles during health care decision making in persons with cancer: a systematic review. Ann Oncol. 2010 Jun;21(6):1145-1151. doi: 10.1093/annonc/mdp534. Epub 2009 Nov 25. PMID 19940010
- [Background] Moth E, McLachlan SA, Veillard AS, Muljadi N, Hudson M, Stockler MR, Blinman P. Patients' preferred and perceived roles in making decisions about adjuvant chemotherapy for non-small-cell lung cancer. Lung Cancer. 2016 May;95:8-14. doi: 10.1016/j.lungcan.2016.02.009. Epub 2016 Feb 21. PMID 27040845
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Padilla-Garrido N, Aguado-Correa F, Ortega-Moreno M, Bayo-Calero J, Bayo-Lozano E. [Shared decision making from the perspective of the cancer patient: participatory roles and evaluation of the process]. An Sist Sanit Navar. 2017 Apr 30;40(1):25-33. doi: 10.23938/ASSN.0003. Spanish. PMID 28534548
- [Derived] Nwachokor J, Rochlin EK, Gevelinger M, Yadav M, Adams W, Fitzgerald C, Acevedo-Alvarez M, Mueller ER, Pham TT. Physician awareness of patients' preferred level of involvement in decision-making at the initial urogynecology visit: a randomized trial. Am J Obstet Gynecol. 2024 Jan;230(1):81.e1-81.e9. doi: 10.1016/j.ajog.2023.06.024. Epub 2023 Jun 15. PMID 37330125